CLINICAL TRIAL: NCT02506036
Title: Efficacy of Web-Based Social-Cognitive Interventions in Right Hemisphere Stroke and Frontotemporal Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061812
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Frontotemporal Dementia; Right Sided Cerebral Hemisphere Cerebrovascular Accident
Keywords: Treatment; Social-Cognitive Training; Web-based; Right Hemisphere Stroke; Frontotemporal Dementia; Right Sided Cerebral Hemisphere Cerebrovascular Accident
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control then Social Cognitive Training (Active Comparator): Patients assigned to this arm will first receive a control therapy on a laptop followed by the Brain HQ social-cognitive training.
  Interventions: Other: Brain HQ
- Social Cognitive Training then Control (Experimental): Patients assigned to this arm will first receive the Brain HQ social-cognitive training and then undergo a control therapy.
  Interventions: Other: Brain HQ

INTERVENTIONS:
Other: Brain HQ — Brain HQ is a web application that will be used to provide patients with a training intervention that addresses deficits in social-emotional functions. These include areas such as identifying facial expression, understanding tone of voice, and predicting how people may react in certain situations. The training will take about 30 hours over the course of 4-6 weeks and is done at home.

SUMMARY:
This study is being done to test the feasibility and effectiveness of web-based social-cognitive training exercises in treating social-emotional deficits in patients with stroke or frontotemporal dementia (FTD).

DETAILED DESCRIPTION:
Although deficits in empathy and social interaction are relatively common in certain forms of FTD and stroke, there are currently no proven treatments for these symptoms. Spouses and caregivers often cite these symptoms as a major concern, and these deficits can have a negative impact on the quality of life that patients experience. The purpose of this study is to evaluate whether or not web-based social training exercises can improve social-cognitive impairments in patients with FTD or right hemisphere stroke. These training exercises have been shown to improve social skills and empathy in other disorders. This study will be the first to examine if these exercises can be effective and feasible for treating social deficits in stroke and FTD.

The study will be based out of the Johns Hopkins Hospital where patients will be assessed three times in total. Patients will be assessed upon enrollment in the study and after each of the two treatment conditions. The training itself will be completed at home on a provided laptop, with monitoring and support by the study team. This study uses a crossover design, which means that all patients will receive the training treatment and a control treatment during their participation in the study. The approximate timeline for the study is 9 weeks total.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of right hemispheric stroke or behavioral variant frontotemporal dementia.
* Able to give informed consent.
* Premorbid proficiency in English (by self-report).
* Age 18 or older.
* Score of 21 or higher on the mini-mental state examination.

Exclusion Criteria:

* Prior history of neurological disease affecting the brain other than stroke or frontotemporal dementia (e.g., brain tumor, multiple sclerosis, traumatic brain injury)
* Known uncorrected hearing loss
* Known uncorrected vision loss
* Prior history of severe psychiatric illness, developmental disorders, or mental retardation (e.g., schizophrenia, autism spectrum disorders) other than FTD
* Score of 20 or lower on the Mini-Mental State Examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argye Hillis, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hosptial, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (4-6 Weeks)
Arm/Group | Control Then Social Cognitive Training | Social Cognitive Training Then Control
Started | 3 | 3
Completed | 2 | 1
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (1-2 Weeks)
Arm/Group | Control Then Social Cognitive Training | Social Cognitive Training Then Control
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Second Intervention (4-6 Weeks)
Arm/Group | Control Then Social Cognitive Training | Social Cognitive Training Then Control
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Then Social Cognitive Training | Social Cognitive Training Then Control | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66.7 [62 to 73] | 67.3 [61 to 73] | 67 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6
Number of Stars Missed On Star Cancellation Test [Median (Full Range); unit: Number of Stars Not Cancelled] — Participants circle every star on a page, in which stars are intermixed with other figures. There are a total of 54 stars. The score is the number of stars that the participant failed to circle. A low number of stars missed (eg. 1 or 2 out of a total of 54) indicates no major visual impairment given then they were able to see and circle almost all of the stars.
  Number of Stars Not Cancelled | 1 [0 to 2] | 1 [0 to 1] | 1 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Social-Cognitive Functioning
Description: Participants will be administered a test of facial emotion recognition called the Penn Emotion recognition task (Range of Scores: 0-40). Participants are shown a face and asked to identify the emotion the face displays, if any. The score reflects the number of faces where the emotion is correctly identified. A score of 35 means that the emotions of 35 out of the 40 faces was correctly identified.
Time Frame: Baseline, after intervention (4 - 6 weeks)
Measure: Mean (Full Range); unit: Number Correct
Groups:
- Social Cognitive Training: This is a combined group of all patients who completed social cognitive training during the study regardless of whether they completed the control condition first or second. The scores reported were taken before and immediately after completion of the training intervention specifically.
  Brain HQ: Brain HQ is a web application that will be used to provide patients with a training intervention that addresses deficits in social-emotional functions. These include areas such as identifying facial expression, understanding tone of voice, and predicting how people may react in certain situations. The training will take about 30 hours over the course of 4-6 weeks and is done at home.
- Control: This is a combined group of all patients who received the control condition and who completed all testing. The scores reported were taken before and immediately after completion of the control portion specifically.
  Control: Participants were given an comparable amount (35 hours) of audiobooks to listen to at home over a 4-6 week period.
Arm/Group | Social Cognitive Training | Control
Number analyzed (Participants) | 3 | 3
Number Correct
  Facial Emotion Recognition At Baseline | 34.6 [34 to 36] | 34.6 [34 to 36]
  Facial Emotion Recognition After Intervention | 35.3 [34 to 38] | 34.6 [34 to 36]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of participation in the study, which on average was between 12-14 weeks dependent on patient availability for testing.
Groups:
- Social Cognitive Training: This is a combined group of all patients who received social cognitive training during the study regardless of whether they completed the control condition first or second. This includes patients who did not finish the training but started it.
  Brain HQ: Brain HQ is a web application that will be used to provide patients with a training intervention that addresses deficits in social-emotional functions. These include areas such as identifying facial expression, understanding tone of voice, and predicting how people may react in certain situations. The training will take about 30 hours over the course of 4-6 weeks and is done at home.
- Control: This is a combined group of all patients who received the control condition during the study. This includes patients who did not finish the control condition but started it.
  Control: Participants were given an comparable amount (35 hours) of audiobooks to listen to at home over a 4-6 week period.
Arm/Group | Social Cognitive Training | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
This was a small scale feasibility study mainly designed to determine how this kind of computerized treatment can be tailored for patients with either frontotemporal dementia or right hemisphere stroke. Further trials will be needed to test efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT02506036/Prot_SAP_000.pdf